CLINICAL TRIAL: NCT04327596
Title: Randomized Clinical Trial of Radiofrequency Ablation for Atrial Fibrillation in Patients With Heart Failure With Preserved Ejection Fraction for Reduced Healthcare Utilization
Brief Title: Radiofrequency (RF) Ablation for Atrial Fibrillation (AF) in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: AF-HFpEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of Rochester (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Mehmet Aktas, Professor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00004367
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Subjects will undergo early RF ablation of AF using CARTO 3 and a Thermocool ST SF ablation catheter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (No Intervention): Subjects will receive management of AF consisting of either rate or rhythm control.
- AF Ablation (Active Comparator): Subjects will undergo early RF ablation of AF using CARTO 3 and a Thermocool ST SF ablation catheter
  Interventions: Procedure: RF ablation of AF using CARTO 3 and a Thermocool ST SF ablation catheter

INTERVENTIONS:
Procedure: RF ablation of AF using CARTO 3 and a Thermocool ST SF ablation catheter — Ablation of AF is standard of care in the management of patients with paroxysmal or persistent AF. The most common triggers initiating AF arise from pulmonary veins (PV) and successful electrical isolation of PV's can significantly reduce the burden of AF. Therefore, the main objective in patients undergoing ablation of AF is to achieve PV isolation.
  Arms: AF Ablation

SUMMARY:
The purpose of this study is to determine if patients who receive an early radiofrequency ablation will have fewer hospitalizations, unplanned office visits, and emergency room visits than those patients treated with medical therapy alone.

DETAILED DESCRIPTION:
In this study, subjects with HFpEF and new onset paroxysmal or persistent AF (diagnosed in the past 6 months) will be randomized in a 1:1 ratio to either intervention or medical therapy alone. Twenty subjects will be enrolled to each group for a total of 40 subjects across all enrolling sites. Subjects randomized to the intervention Group will undergo early RF ablation of AF using CARTO 3 and a Thermocool ST SF ablation catheter. The medical therapy alone cohort will receive management of AF consisting of either rate or rhythm control. All patients will be implanted with an implantable cardiac monitor (ICM) as standard of care for AF management in heart failure except for those who already have in place an existing cardiac implantable electronic device (CIED) such as pacemaker, ICM, or implantable cardiac defibrillator (ICD). The ICM procedure will occur within 2 calendar months of randomization for both study groups (intervention or control). For the intervention arm, the CIED procedure will occur prior to or at the time of the AF ablation procedure. Subjects will be followed for 1 year with in-clinic visits occurring at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years at date of consent.
* LVEF >50% as determined on imaging study measured in the last 6 calendar months prior to or on consent date.
* Hospitalized for HF within the past 12 calendar months prior to consent date.
* Stabilized patients defined as being off all IV therapies for at least 24 hours prior to consent date.
* Paroxysmal AF diagnosed within the past 6 calendar months or early persistent AF, defined as an AF episode lasting greater than 7 days but less than 6 calendar months prior to consent date.
* Indicated for oral anticoagulation according to current guidelines (CHA2DS2-VASc ≥ 2 in men or ≥ 3 in women at the time of consent)*
* Patient with CIED in situ at time of consent or scheduled to undergo ICM implant for AF management within 2 calendar months of randomization.

Exclusion Criteria:

* Previous catheter or surgical ablation of AF any time in the past.
* Long-standing persistent AF (>1-year prior to consent date) or permanent AF.
* Chronic pulmonary disease requiring home oxygen or oral/IV steroid therapy in the past 12 calendar months prior to consent date.
* Active infection at time of consent but may be re-considered for enrollment later after effective treatment.
* Left atrial size >50 mm as measured by echo in the past 6 calendar months prior to consent date.
* Untreated obstructive sleep apnea any time in past.
* Myocardial infarction in past 3 calendar months prior to consent date.
* Coronary artery bypass graft (CABG) surgery in past 3 calendar months prior to consent date.
* Stroke in past 3 calendar months prior to consent date.
* Intra-cardiac thrombus precluding ability to undergo AF ablation at time of consent but may be re-considered for enrollment later after effective treatment.
* Infiltrative cardiomyopathy (sarcoid, amyloid) any time in past.
* Active myocarditis at time of consent but may be re-considered for enrollment later after effective treatment.
* Hypertrophic cardiomyopathy at any time in past.
* Known pericardial constriction.
* Uncontrolled hypertension (SBP > 160 mmHg) at time of consent but may be re- considered for enrollment later after effective treatment.
* Untreated hypothyroidism or hyperthyroidism but may be re-considered for enrollment later after effective treatment.
* Pregnancy or nursing.
* Valvular AF or presence of a prosthetic valve.
* Undergoing dialysis or have advanced renal dysfunction (eGFR <30 ml/min/m2) defined as 3 times the upper limits of AST or ALT during the past 6 calendar months.
* Contraindication to anticoagulation.
* Metabolic derangements (e.g. renal/hepatic failure, electrolyte disturbance, etc.), prohibiting study (EP) study and ablation.
* Cognitive impairment.
* Life expectancy < 1 year following consent date.
* Unwilling to comply with all study protocol-required testing.
* Unwilling or unable to give informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Rate of healthcare utilization. | up to 12 months
  Number of unplanned office visits, hospitalizations, and emergency room visits.

SECONDARY OUTCOMES:
Burden of Atrial Fibrillation (AF) | Between baseline and 12 months
  Percentage of time spent in AF (i.e. amount of time spent in AF divided by the total amount of CIED monitoring time).
Change in quality of life measures in Patient-Reported Outcomes Measurement Information System (PROMIS). | Between baseline and 6 months
  Consists of 24 questions with a scale of 1-5 with 1 being the worst
6-minute Walk Test | 6 Months
  Mean changes in functional status
Quality of life measures using the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Between baseline and 6 months
  Consists of 8 questions with a scale of 1-5 with 1 being the worst

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K Aktas, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Rochester Regional Health, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] Loehr LR, Rosamond WD, Chang PP, Folsom AR, Chambless LE. Heart failure incidence and survival (from the Atherosclerosis Risk in Communities study). Am J Cardiol. 2008 Apr 1;101(7):1016-22. doi: 10.1016/j.amjcard.2007.11.061. Epub 2008 Feb 14. PMID 18359324
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Kotecha D, Lam CS, Van Veldhuisen DJ, Van Gelder IC, Voors AA, Rienstra M. Heart Failure With Preserved Ejection Fraction and Atrial Fibrillation: Vicious Twins. J Am Coll Cardiol. 2016 Nov 15;68(20):2217-2228. doi: 10.1016/j.jacc.2016.08.048. PMID 27855811
- [Background] Packer M, Colucci WS, Sackner-Bernstein JD, Liang CS, Goldscher DA, Freeman I, Kukin ML, Kinhal V, Udelson JE, Klapholz M, Gottlieb SS, Pearle D, Cody RJ, Gregory JJ, Kantrowitz NE, LeJemtel TH, Young ST, Lukas MA, Shusterman NH. Double-blind, placebo-controlled study of the effects of carvedilol in patients with moderate to severe heart failure. The PRECISE Trial. Prospective Randomized Evaluation of Carvedilol on Symptoms and Exercise. Circulation. 1996 Dec 1;94(11):2793-9. doi: 10.1161/01.cir.94.11.2793. PMID 8941104
- [Background] CONSENSUS Trial Study Group. Effects of enalapril on mortality in severe congestive heart failure. Results of the Cooperative North Scandinavian Enalapril Survival Study (CONSENSUS). N Engl J Med. 1987 Jun 4;316(23):1429-35. doi: 10.1056/NEJM198706043162301. PMID 2883575
- [Background] Cohn JN, Tognoni G; Valsartan Heart Failure Trial Investigators. A randomized trial of the angiotensin-receptor blocker valsartan in chronic heart failure. N Engl J Med. 2001 Dec 6;345(23):1667-75. doi: 10.1056/NEJMoa010713. PMID 11759645
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Background] Cleland JG, Tendera M, Adamus J, Freemantle N, Polonski L, Taylor J; PEP-CHF Investigators. The perindopril in elderly people with chronic heart failure (PEP-CHF) study. Eur Heart J. 2006 Oct;27(19):2338-45. doi: 10.1093/eurheartj/ehl250. Epub 2006 Sep 8. PMID 16963472
- [Background] Pitt B, Pfeffer MA, Assmann SF, Boineau R, Anand IS, Claggett B, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Harty B, Heitner JF, Kenwood CT, Lewis EF, O'Meara E, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, Yang S, McKinlay SM; TOPCAT Investigators. Spironolactone for heart failure with preserved ejection fraction. N Engl J Med. 2014 Apr 10;370(15):1383-92. doi: 10.1056/NEJMoa1313731. PMID 24716680
- [Background] Yamamoto K, Origasa H, Hori M; J-DHF Investigators. Effects of carvedilol on heart failure with preserved ejection fraction: the Japanese Diastolic Heart Failure Study (J-DHF). Eur J Heart Fail. 2013 Jan;15(1):110-8. doi: 10.1093/eurjhf/hfs141. Epub 2012 Sep 14. PMID 22983988
- [Background] Yusuf S, Pfeffer MA, Swedberg K, Granger CB, Held P, McMurray JJ, Michelson EL, Olofsson B, Ostergren J; CHARM Investigators and Committees. Effects of candesartan in patients with chronic heart failure and preserved left-ventricular ejection fraction: the CHARM-Preserved Trial. Lancet. 2003 Sep 6;362(9386):777-81. doi: 10.1016/S0140-6736(03)14285-7. PMID 13678871
- [Background] Santhanakrishnan R, Wang N, Larson MG, Magnani JW, McManus DD, Lubitz SA, Ellinor PT, Cheng S, Vasan RS, Lee DS, Wang TJ, Levy D, Benjamin EJ, Ho JE. Atrial Fibrillation Begets Heart Failure and Vice Versa: Temporal Associations and Differences in Preserved Versus Reduced Ejection Fraction. Circulation. 2016 Feb 2;133(5):484-92. doi: 10.1161/CIRCULATIONAHA.115.018614. Epub 2016 Jan 8. PMID 26746177
- [Background] Goyal P, Almarzooq ZI, Cheung J, Kamel H, Krishnan U, Feldman DN, Horn EM, Kim LK. Atrial fibrillation and heart failure with preserved ejection fraction: Insights on a unique clinical phenotype from a nationally-representative United States cohort. Int J Cardiol. 2018 Sep 1;266:112-118. doi: 10.1016/j.ijcard.2018.02.007. PMID 29887426
- [Background] Cikes M, Claggett B, Shah AM, Desai AS, Lewis EF, Shah SJ, Anand IS, O'Meara E, Rouleau JL, Sweitzer NK, Fang JC, Saksena S, Pitt B, Pfeffer MA, Solomon SD. Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction: The TOPCAT Trial. JACC Heart Fail. 2018 Aug;6(8):689-697. doi: 10.1016/j.jchf.2018.05.005. Epub 2018 Jul 11. PMID 30007557
- [Background] Zakeri R, Chamberlain AM, Roger VL, Redfield MM. Temporal relationship and prognostic significance of atrial fibrillation in heart failure patients with preserved ejection fraction: a community-based study. Circulation. 2013 Sep 3;128(10):1085-93. doi: 10.1161/CIRCULATIONAHA.113.001475. Epub 2013 Aug 1. PMID 23908348
- [Background] Rosenberg MA, Gottdiener JS, Heckbert SR, Mukamal KJ. Echocardiographic diastolic parameters and risk of atrial fibrillation: the Cardiovascular Health Study. Eur Heart J. 2012 Apr;33(7):904-12. doi: 10.1093/eurheartj/ehr378. Epub 2011 Oct 11. PMID 21990265
- [Background] Tsang TS, Gersh BJ, Appleton CP, Tajik AJ, Barnes ME, Bailey KR, Oh JK, Leibson C, Montgomery SC, Seward JB. Left ventricular diastolic dysfunction as a predictor of the first diagnosed nonvalvular atrial fibrillation in 840 elderly men and women. J Am Coll Cardiol. 2002 Nov 6;40(9):1636-44. doi: 10.1016/s0735-1097(02)02373-2. PMID 12427417
- [Background] Oluleye OW, Rector TS, Win S, McMurray JJ, Zile MR, Komajda M, McKelvie RS, Massie B, Carson PE, Anand IS. History of atrial fibrillation as a risk factor in patients with heart failure and preserved ejection fraction. Circ Heart Fail. 2014 Nov;7(6):960-6. doi: 10.1161/CIRCHEARTFAILURE.114.001523. Epub 2014 Sep 15. PMID 25225241
- [Background] Sartipy U, Dahlstrom U, Fu M, Lund LH. Atrial Fibrillation in Heart Failure With Preserved, Mid-Range, and Reduced Ejection Fraction. JACC Heart Fail. 2017 Aug;5(8):565-574. doi: 10.1016/j.jchf.2017.05.001. Epub 2017 Jul 12. PMID 28711451
- [Background] Nattel S, Harada M. Atrial remodeling and atrial fibrillation: recent advances and translational perspectives. J Am Coll Cardiol. 2014 Jun 10;63(22):2335-45. doi: 10.1016/j.jacc.2014.02.555. Epub 2014 Mar 19. PMID 24613319
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Joseph SM, Novak E, Arnold SV, Jones PG, Khattak H, Platts AE, Davila-Roman VG, Mann DL, Spertus JA. Comparable performance of the Kansas City Cardiomyopathy Questionnaire in patients with heart failure with preserved and reduced ejection fraction. Circ Heart Fail. 2013 Nov;6(6):1139-46. doi: 10.1161/CIRCHEARTFAILURE.113.000359. Epub 2013 Oct 15. PMID 24130003
- [Background] Yee D, Novak E, Platts A, Nassif ME, LaRue SJ, Vader JM. Comparison of the Kansas City Cardiomyopathy Questionnaire and Minnesota Living With Heart Failure Questionnaire in Predicting Heart Failure Outcomes. Am J Cardiol. 2019 Mar 1;123(5):807-812. doi: 10.1016/j.amjcard.2018.11.037. Epub 2018 Dec 4. PMID 30587373
- [Background] Napier R, McNulty SE, Eton DT, Redfield MM, AbouEzzeddine O, Dunlay SM. Comparing Measures to Assess Health-Related Quality of Life in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2018 Jul;6(7):552-560. doi: 10.1016/j.jchf.2018.02.006. Epub 2018 Jun 6. PMID 29885952
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Bruckel J, Wagle N, O'Brien C, Elias J, McKenna S, Meyers P, Fifer MA, Pomerantsev E, Yeh RW. Feasibility of a Tablet Computer System to Collect Patient-reported Symptom Severity in Patients Undergoing Diagnostic Coronary Angiography. Crit Pathw Cardiol. 2015 Dec;14(4):139-45. doi: 10.1097/HPC.0000000000000058. PMID 26569653
- [Background] Nattel S, Guasch E, Savelieva I, Cosio FG, Valverde I, Halperin JL, Conroy JM, Al-Khatib SM, Hess PL, Kirchhof P, De Bono J, Lip GY, Banerjee A, Ruskin J, Blendea D, Camm AJ. Early management of atrial fibrillation to prevent cardiovascular complications. Eur Heart J. 2014 Jun 7;35(22):1448-56. doi: 10.1093/eurheartj/ehu028. Epub 2014 Feb 16. PMID 24536084
- [Background] Marrouche NF, Brachmann J, Andresen D, Siebels J, Boersma L, Jordaens L, Merkely B, Pokushalov E, Sanders P, Proff J, Schunkert H, Christ H, Vogt J, Bansch D; CASTLE-AF Investigators. Catheter Ablation for Atrial Fibrillation with Heart Failure. N Engl J Med. 2018 Feb 1;378(5):417-427. doi: 10.1056/NEJMoa1707855. PMID 29385358
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041